CLINICAL TRIAL: NCT05591391
Title: The Efficacy of Mallya in Type 2 Diabetes Transiting From Oral Antidiabetic Drugs to iGlarLixi: a Randomized Controlled Trial Using Real-time Continuous Glucose Monitoring
Brief Title: The Efficacy of Mallya in Type 2 Diabetes Transiting From Oral Antidiabetic Drugs to iGlarLixi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Attetnding Physician, Department of Endocrinology and Metabolism, Principal Investigator, Doctor of Philosophy, Associate Professor, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-07-010B
Record Dates: First submitted 2022-10-02; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Mallya
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mallya (Experimental): Patients use Mallya cap to record the time and dosage of insulin injection
  Interventions: Other: Mallya cap
- Standard care (Active Comparator): Patients receive standard care.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Mallya cap — After Mallya cap is correctly attached to the insulin pen, it will automatically record treatment information (dose, time and date of injection) and send in real time to the Health2Sync's platform by Bluetooth transmission. Suggestions regarding dose titration and glycemic control will be communicated on the Health2Sync's platform.
  Arms: Mallya
Other: Standard care — Suggestions regarding dose titration and glycemic control will be communicated by weekly telephone calls.
  Arms: Standard care

SUMMARY:
This is a randomized, 12-week, open-label, active-controlled, parallel group study that will collect data of real-time continuous glucose monitoring for seven days at baseline and the end of study from adults with Type 2 diabetes mellitus inadequately controlled on oral antidiabetic drugs transiting to their first injectable therapy, iGlarLixi. A total of 40 patients will be recruited in Taipei Veterans General Hospital and randomized to use Mallya or receive standard care. The study is designed to demonstrate the efficacy of Mallya compared to standard care in terms of time in range (glucose level of 70-180 mg/dL), time above range (glucose level ≥180 mg/dL), time below range (glucose level <70 mg/dL), glycemic variability indices, changes in HbA1c and percentage of patients with HbA1c ≤7.0% at endpoint, time to stable dose, and diabetes treatment satisfaction. The result of the current study will provide insights into the utility of Mallya as a treatment monitoring solution to improve glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years-old
* T2DM ≥ 180 days
* HbA1c ≥ 7.0% at screening
* Under stable doses of OADs for ≥12 weeks prior to screening
* Insulin naïve (except short term insulin treatment for a maximum of 14 days before screening and/or prior insulin treatment for gestational diabetes)
* Not currently using real time continuous or flash glucose monitoring
* Not currently using Mallya

Exclusion Criteria:

* Known or suspected hypersensitivity to randomized treatment or related products
* Previous participation in this study (Participation is defined as signed informed consent);
* Participation (i.e., signed informed consent) in any interventional, clinical study within 90 days before screening (except for COVID-19 study);
* Female who is pregnant, breast-feeding or intends to become pregnant
* Presence of severe gastrointestinal disorders, such as severe gastroparesis;
* Presence of severe renal dysfunction (eGFR <30 ml/min/1.73 m2) or end-stage renal disease on dialysis;
* Presence of severe hepatic dysfunction (AST or ALT level ≥ 200 U/L);
* Patients with a history of pancreatitis;
* Patients receiving systemic corticosteroids
* Patients with active cancer within the past six months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Time in range | 7 days of CGM data
  The time in range (TIR) in percent (%) of a glucose level of 70-180 mg/dL obtained by real-time continuous glucose monitoring (rt-CGM) at the end of the study in both groups.

SECONDARY OUTCOMES:
Time above range (TAR) | 7 days of CGM data
  Time above range (TAR) in percent (%) of a glucose level ≥180 mg/dL
Time below range (TBR) | 7 days of CGM data
  Time below range (TBR) in percent (%) of a glucose level <70 mg/dL and nocturnal (00.00-06.00 hours) TBR
Mean of glucose levels | 7 days of CGM data
  Mean in mg/dL of glucose levels obtained on rt-CGM
Standard deviation (SD) of glucose levels | 7 days of CGM data
  Standard deviation (SD) in mg/dL of glucose levels obtained on rt-CGM
Coefﬁcient of variation (CV) of glucose levels | 7 days of CGM data
  Coefﬁcient of variation (CV) in mg/dL of glucose levels obtained on rt-CGM
HbA1c | 12 weeks
  Changes in HbA1C (post-study HbA1C minus pre-study HbA1C) and percentage of patients with HbA1C ≤7.0%
Time to stable dose | 12 weeks
  The time (days) for patients to achieve target fasting glucose level and stable dose of iGlarLixiThe
Treatment satisfaction questionnaire | 12 weeks
  Diabetes Treatment Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology and Metabolism, Department of Medicine, Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No